CLINICAL TRIAL: NCT03823612
Title: Reminerlization Potential of Innovative Biomimetic Material Versus Casein Phosphopeptide-amorphous Calcium Phosphate in Caries White Spot Lesions "A Randomized Clinical Trial"
Brief Title: Reminerlization Potential of Innovative Biomimetic Material in Caries White Spot Lesions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, donia mahmoud abd el moaty; Doniamahmoud17@gmail.com, principle investigator in cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: donia mahmoud
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: White Spot Lesion of Tooth
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC tooth mousse (Experimental): Drug: GC tooth mousse it contains complex of Casein Phosphopeptide,Amorphous Calcium Phosphate ( CPP-ACP ) other name: Tooth Mousse (Bio-available calcium and phosphate, without fluoride)
  Interventions: Drug: GC tooth mousse
- clinpro tooth creme (Active Comparator): it contains 0.21% Sodium Fluoride, Anti-Cavity Paste is an advanced formula containing an innovative tri-calcium phosphate ingredient
  other name:0.21% w/w Sodium Fluoride Anti-Cavity Paste with Tri-Calcium Phosphate
  Interventions: Drug: Clinpro Tooth Creme

INTERVENTIONS:
Drug: Clinpro Tooth Creme — The participant will be instructed to Place a pea-sized amount of Clinpro Tooth Crème on a soft bristled toothbrush and brush teeth for at least two minutes then after brushing the patient will rinse out his mouth with water and spit out. It will be used twice daily at first in the morning and before sleep.
  Other Names: Anti-Cavity Paste with Tri-Calcium Phosphate
  Arms: clinpro tooth creme
Drug: GC tooth mousse — The participant will be instructed to squeeze a small amount of GC Tooth Mousse out onto a clean finger. A cotton tip, swab or custom tray are suitable application methods as it will Applied directly onto his tooth surfaces and leave undisturbed for three minutes then he will be instructed to Spread any residual crème around the mouth with his tongue and hold for a further one to two minutes then the participant will expectorate thoroughly and if possible he should avoid rinsing. Any GC Tooth Mousse remaining in the mouth can be left to gradually dissipate. The participant will be instructed to avoid eating or drinking for 30 minutes following application.
  Arms: GC tooth mousse

SUMMARY:
to remineralize the white spot caries lesions after orthodontic treatment , the investigator will use two different materials ( Clinpro tooth creme versus Gc tooth mousse) and will compare between their effects in remineralization of white spot caries lesions.

DETAILED DESCRIPTION:
Dental caries is the localized destruction of tooth tissues by acids, especially lactic acid, produced by the fermentation of dietary carbohydrates by bacteria in dental plaque. Demineralization can be arrested or reversed when remineralization agents are applied to incipient carious or non-cavitated carious lesions. A large number of therapeutic agents including non-fluoridated products have been developed to promote enamel remineralization. The process of restoring lost mineral ions to the tooth structure and strengthening the lattice work is known as remineralization.

The development of decalcification around orthodontic brackets and bands, commonly called white spot lesions (WSLs), is often observed in patients with poor oral hygiene during treatment .In many instances, these WSLs continue to be visible after the removal of fixed appliances and after natural remineralization. The remineralized enamel crystallites are generally more resistant to decalcification and also have the same orientation as the original enamel crystallites. The early enamel lesions have a potential for remineralization with an increased resistance to further acid challenge, particularly with the use of enhanced remineralization treatments.

Recaldent™ is derived from the milk protein, casein. For many years it has been known that milk and its derivatives have a tooth protective effect. Research has shown that this activity is due to a part of the casein protein called Casein Phosphopeptide (or CPP), which carries calcium and phosphate ions in the form of Amorphous Calcium Phosphate (or ACP) which used in reminerlization of white spot caries lesions.

Clinpro tooth crème (3M ESPE) is a 0.21% w/w sodium fluoride (NaF) anti caries dentifrice that contains 950 ppm fluoride and a functionalized tricalcium phosphate (f-TCP) ingredient.One major advantage of this calcium phosphate system is that it is stable in aqueous environment and also does not affect the fluoride activity added in the dentifrices. Furthermore,it has been suggested that fluoride combination with f-TCP not only provides greater remineralization in terms of microhardness and fluoride uptake, but also decreases the dose of fluoride required to achieve the same degree of remineralization,

ELIGIBILITY:
Inclusion Criteria:

* Patients should have at least one white spot caries lesion
* age from 18 to 40 years
* no gender restriction

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease
* Patients with developmental hypo-calcified lesions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
esthetic assessment | baseline, after 1 month , 3 months and 6 months of the application
  Spectrophotometer ( L, a, b) will be used to measure the change in the shade of the white spot lesions during the study

SECONDARY OUTCOMES:
patient compliance | 6 months
  The participants compliance will be detected by a questionnaire by asking the patient to describe his satisfaction to the total outcome of our intervention by giving a score from 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Donia Mahmoud Abd El Moaty, Cairo, Egypt